CLINICAL TRIAL: NCT06834256
Title: Intermittent Fasting vs. High-Intensity Interval Training on Lipid Profile in Obese Patients
Brief Title: Intermittent Fasting vs. High-intensity Interval Training on the Lipid Profile of Obese Individuals.
Acronym: vs(versus)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Ahmed Mousa, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004625
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Obesity
Keywords: Intermittent Fasting,High-Intensity Training,,Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (IF group) (Experimental): Group A followed the intermittent fasting( IF) regime ,with an intervention duration of six weeks for both groups
  Interventions: Behavioral: intermittent fasting
- Group B performed High-intensity interval training( HIIT) (Experimental): High-intensity interval training performed on the treadmill three times weekly, with an intervention duration of six weeks for both groups
  Interventions: Behavioral: low volume high intensity interval training

INTERVENTIONS:
Behavioral: intermittent fasting — Group A participants followed the IF diet for 6 weeks . intermittent fasting , specifically time-restricted feeding (TRF), involves consuming all of one's energy requirements inside an 8-h.The fasting interval was designated as 16 h, and the other 8-h was the eating period . During the 8-h eating window, the patient consumes a well-balanced meal consisting of 55%-65% carbs, 7%-20% protein, and 15%-30% fat .
  Arms: Group A (IF group)
Behavioral: low volume high intensity interval training — . Group B engaged in low-volume HIIT exercise (aerobic activity) three times weekly for six weeks. The exercise routine consisted of a 5-min warm-up phase at 70% of MHR, followed by four intervals of 2-min maximum effort cycling sessions (4 × 2 HIIT) compared to a sub-maximal workload at 85%-90% of MHR. The participants engaged in four work bouts, with each bout lasting around 4 min and followed by a 4-min rest period. During the workouts, the participants maintained an HR of 60%-70% of their MHR. This resulted in 8 min of intense physical activity during each training session. Additionally, there was a 5-min cooling down phase at 70% of the MHR. The treatment's intensity was adapted based on the modified Bruce protocol.
  Arms: Group B performed High-intensity interval training( HIIT)

SUMMARY:
we aimed to ascertain the effect of intermittent fasting (IF) vs. high-intensity interval training (HIIT) on the lipid profile and waist circumference (WC) of obese individuals.

DETAILED DESCRIPTION:
Subjects and Methods: This study included 40 obese individuals of both genders aged 35-50 years with an abnormal lipid profile. The patients were allocated at random to either Group A or B, with both groups receiving medical treatment. Group A followed the IF regime, while Group B performed HIIT on the treadmill three times weekly, with an intervention duration of six weeks for both groups. Body mass index (BMI), WC, levels of total cholesterol (TC), triglyceride (TG), low-density lipoprotein (LDL), high-density lipoprotein (HDL), alongside the Framingham risk score (FRS) were the evaluated variables.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were as follows: (1) A BMI of 30 -40 kg/m2; (2) abnormal lipid profile, with a TC level > 200 mg/dL, an LDL > 100 mg/dL, a TC level > 150 mg/dL, and an HDL < 40 mg/dL; (3) steady vital signs, including blood pressure, respiration rate, and temperature at a baseline level.

Exclusion Criteria:

* The exclusion criteria included patients with the following medical conditions: cancer, unstable angina, uncontrolled cardiac rhythm, decompensated heart failure, persistent systolic blood pressure > 200 mmHg, persistent diastolic blood pressure > 120 mmHg, acute pericarditis or myocarditis, severe restrictive lung disease, chronic chest infection, severe obstructive lung disease, pregnant women, neurological disorders that affect balance and mentality (e.g., epilepsy), orthopedic or neurological problems that interfere with exercises, unstable endocrinal disorders, congenital or acquired lower limb deformity, kidney disease, infectious disease, immune disease, hearing impairment or mental disorder, uncontrolled T2DM.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-03-02 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
lipid profile | lipid profile will be measured at baseline, and it will be measured again after six weeks
  A 5 mL fasting venous blood sample was collected following an eight-hour overnight fast, and LDL, HDL, TG, and TC levels were measured.

SECONDARY OUTCOMES:
waist circumference | waist circumference will be measured at baseline, and it will be measured again after six weeks
  Utilizing tape measurements to measure WC.A WC > 40 inches (102 cm) in males and > 35 inches (88 cm) in women indicated an elevated risk for cardiometabolic disorders
The Framingham risk score (FRS) | The Framingham risk score (FRS) will be measured at baseline, and it will be measured again after six weeks
  It was employed to ascertain the cardiovascular disease risk over ten years.

CONTACTS AND LOCATIONS:
Overall Officials: Heba Mousa, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

REFERENCES:
- [Result] Nussbaumerova B, Rosolova H. Obesity and Dyslipidemia. Curr Atheroscler Rep. 2023 Dec;25(12):947-955. doi: 10.1007/s11883-023-01167-2. Epub 2023 Nov 18. PMID 37979064
- [Result] Nazari M, Minasian V, Hovsepian S. Effects of Two Types of Moderate- and High-Intensity Interval Training on Serum Salusin-alpha and Salusin-beta Levels and Lipid Profile in Women with Overweight/Obesity. Diabetes Metab Syndr Obes. 2020 Apr 24;13:1385-1390. doi: 10.2147/DMSO.S248476. eCollection 2020. PMID 32425570